CLINICAL TRIAL: NCT00667472
Title: Combined Pulsed Dye Laser and Topical Ranibizumab for Treatment of Port Wine Stain Birthmarks
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, J.S.Nelson, MD,PhD,Professor of Surgery and Biomedical Engineering, University of California, Irvine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 20076098
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Port-Wine Stain
Keywords: port wine stain birthmarks
MeSH Terms: conditions — Port-Wine Stain | interventions — Ranibizumab; Lasers, Dye

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranibizumab (Experimental): Combined Pulsed Dye Laser and Topical Ranibizumab for Treatment of Port Wine Stain Birthmarks
  Interventions: Drug: Ranibizumab
- Pulsed Dye Laser (Experimental): Combined Pulsed Dye Laser and Topical Ranibizumab for Treatment of Port Wine Stain Birthmarks
  Interventions: Device: Pulsed Dye Laser

INTERVENTIONS:
Drug: Ranibizumab — Combined Pulsed Dye Laser and Topical Ranibizumab for Treatment of Port Wine Stain Birthmarks
  Arms: Ranibizumab
Device: Pulsed Dye Laser — Combined Pulsed Dye Laser and Topical Ranibizumab for Treatment of Port Wine Stain Birthmarks
  Arms: Pulsed Dye Laser

SUMMARY:
The purpose of this study is to improve port wine stain therapeutic outcome in response to laser therapy. The researcher want to determine whether the combined use of pulsed dye laser therapy and topical ranibizumab will improve port wine stain therapeutic outcome.

DETAILED DESCRIPTION:
Combined use of pulsed dye laser to induce port wine stain blood vessel injury, and ranibizumab to prevent port wine stain blood vessel angiogenesis and recanalization after laser therapy, will improve port wine stain lesion blanching.

After pulsed dye laser treatment of the entire port wine stain, topical ranibizumab will be applied to two of the test sites for two weeks following pulsed dye laser therapy. The degree of port wine stain blanching which will be quantified objectively using visible reflectance spectroscopy measurements. port wine stain test site blanching responses following the combined use of pulsed dye laser and topical ranibizumab will be compared with pulsed dye laser only and with the baseline controls.

ELIGIBILITY:
Inclusion Criteria:

* Port Wine Stain suitable for comparison testing
* Age > 18 years of age

Exclusion Criteria:

* History of photodermatoses or skin cancer
* use of known photosensitizing drugs
* use of immunosuppressive drugs or systemic steroids
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Port Wine Stain response to laser treatment | 8 weeks
  Combined Pulsed Dye Laser and Topical Ranibizumab for Treatment of Port Wine Stain Birthmarks

CONTACTS AND LOCATIONS:
Overall Officials: John s Nelson, M.D,PhD, Principal Investigator — Beckman Laser Institute University of California Irvine